## **CONSENT FORM**



Study number:

discussed consent

Participant identification number:

| | • | | | |
|---|---|---|---|---|
| | <b>f Project</b> : An Electronic Patien<br>omized Control Trial | t Decision Aid for | r Antidepressant Use in Pregr | nancy: Pilot |
| Chief | Investigator: Louise M. Howard | | | |
| In order to take part, please confirm that you are happy with the following: | | | | Please<br>tick |
| 1. | I confirm that I have read and understood the Participant Information Sheet [v2, 27/11/2015] for the above study. I have had the opportunity to think about the information, ask questions about the study, and have had my questions answered. | | | |
| 2. | I understand that taking part in the study is voluntary and that I can leave at any time, without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | . I agree to take part in this study. | | | |
| 4. | I give permission for researchers to contact my clinical team (midwife, doctor, nurse) to inform them about the study and check my eligibility to take part. | | | |
| | parts of the study are optional,<br>ing (delete as appropriate): | , please indicate w | hether or not you agree to the | |
| 5. | 5. I give permission for researchers to have access to my medical records for the collection of data that is relevant to this research. | | | YES / NO |
| 6. | I agree to the audiotaping of my first appointment with my doctor after I use the study website. | | | |
| 7. | 7. I agree to be contacted by the researchers about ethically approved related YES / | | | |
| 8. | studies. 8. I would like to be sent a summary of the research findings upon completion of | | | YES / NO |
| Name of participant | | Date | Signature (If consentir type your initials to indicate | |
| | То | be completed by re | esearcher: | |
| Name of researcher who | | Date | Signature | |

When completed: one copy for participants, one copy for researcher site file.

V3, 27/11/2015 1